CLINICAL TRIAL: NCT00386867
Title: A Randomized Trial of Buccal Compared to Oral Misoprostol Following Mifepristone for Medical Abortion up to 63 Days LMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.1.3
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2007-06-05 (Estimated); Status verified 2007-06

CONDITIONS: Abortion, Induced
Keywords: medical abortion; mifepristone; misoprostol; buccal administration
MeSH Terms: interventions — Administration, Buccal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 800 mcg misoprostol via oral or buccal administration

SUMMARY:
This open-label, randomized study will compare the efficacy, safety, and acceptability of mifepristone 200 mg followed in 24-36 hours either by buccal (i.e., in the cheeks) or oral misoprostol 800 mcg for termination of pregnancy in women up to 63 days L.M.P.

ELIGIBILITY:
Inclusion Criteria:

* be willing and able to sign consent forms;
* be eligible for medical abortion according to clinician's assessment;
* be willing to undergo a surgical completion if necessary;
* have ready and easy access to a telephone and emergency transportation;
* speak English, Spanish, or have a translator available to translate for all study procedures; and,
* agree to comply with the study procedures and visit schedule.

Exclusion Criteria:

* Confirmed or suspected ectopic pregnancy or undiagnosed adnexal mass;
* IUD in place;
* Chronic renal failure;
* Concurrent long-term corticosteroid therapy;
* History of allergy to mifepristone, misoprostol or other prostaglandin;
* Hemorrhagic disorders or concurrent anticoagulant therapy;
* Inherited porphyrias; or
* Other serious physical or mental health conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2006-10; Study Completion 2007-03

PRIMARY OUTCOMES:
efficacy

SECONDARY OUTCOMES:
acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Ilana Dzuba, MHS, Study Director — Gynuity Health Projects
Locations (8):
- United States (8):
  - Family Planning Associates Medical Group, Chicago, Illinois
  - Planned Parenthood League of Massachusetts (Boston clinic), Boston, Massachusetts
  - Columbia University Medical Center, Division of Obstetrics & Gynecology, New York, New York
  - Institute for Urban Family Health, New York, New York
  - Parkmed, New York, New York
  - University of Pittsburgh, Division of Obstetrics, Gynecology and Reproductive Sciences, Pittsburgh, Pennsylvania
  - Whole Women's Health, Austin, Texas
  - Planned Parenthood, Waco, Texas

REFERENCES:
- [Derived] Winikoff B, Dzuba IG, Creinin MD, Crowden WA, Goldberg AB, Gonzales J, Howe M, Moskowitz J, Prine L, Shannon CS. Two distinct oral routes of misoprostol in mifepristone medical abortion: a randomized controlled trial. Obstet Gynecol. 2008 Dec;112(6):1303-1310. doi: 10.1097/AOG.0b013e31818d8eb4. PMID 19037040
- See also: Related Info — http://www.gynuity.org